CLINICAL TRIAL: NCT04790864
Title: Speaking Out Against Anxiety: Feasibility and Efficacy of an Online Large-group One-session Treatment for Public Speaking Anxiety and the Role of Expectancy Violation
Brief Title: An Online Large-group One-session Treatment for Public Speaking Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Svenja Schaumburg, Principal Investigator (Research Fellow / PhD Student), Ruhr University of Bochum
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 684
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Anxiety, Social
Keywords: large-group treatment; one-session treatment; online intervention; public speaking anxiety; expectancy violation
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants are not aware that there are two different post-treatment exercises and are not informed that the aim of the EV condition is to promote expectancy violation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online large-group one-session treatment with post-treatment exercise targeting expectancy violation (Experimental)
  Interventions: Behavioral: Online large-group one-session treatment with post-treatment exercise targeting expectancy violation
- Online large-group one-session treatment with post-treatment control exercise (Active Comparator)
  Interventions: Behavioral: Online large-group one-session treatment with post-treatment control exercise

INTERVENTIONS:
Behavioral: Online large-group one-session treatment with post-treatment exercise targeting expectancy violation — The treatment is aimed at reducing public speaking anxiety by using cognitive and behavioral techniques. Following a psychoeducation phase, different speaking tasks are conducted to expose the individuals to their feared situation on the one hand and to address common cognitive processes characterizing public speaking anxiety, e.g. self-focused attention, on the other hand. The exercises will be conducted in smaller groups. After treatment, participants receive a worksheet with questions aimed at enhancing the processing of what was learned during treatment in terms of expectancy violation. For example, they are asked if what they were most worried about occured and what actually happened compared to what they predicted to happen. This should highlight the discrepancy between anticipated and actual outcomes. The intervention is conducted in an online group format via videoconference with a duration of approximately 5 hours.
  Arms: Online large-group one-session treatment with post-treatment exercise targeting expectancy violation
Behavioral: Online large-group one-session treatment with post-treatment control exercise — The treatment is aimed at reducing public speaking anxiety by using cognitive and behavioral techniques. Following a psychoeducation phase, different speaking tasks are conducted to expose the individuals to their feared situation on the one hand and to address common cognitive processes characterizing public speaking anxiety, e.g. self-focused attention, on the other hand. The exercises will be conducted in smaller groups. After treatment, participants receive a worksheet that addresses basic contentual information concerning the treatment without a specific attempt to highlight the discrepancy between anticipated and actual outcomes. For example, participants will be asked how they would explain public speaking anxiety and exposure therapy to a friend and what advantages they see in conducting treatments like this in groups. The intervention is conducted in an online group format via videoconference with a duration of approximately 5 hours.
  Arms: Online large-group one-session treatment with post-treatment control exercise

SUMMARY:
Different conceptualizations of public speaking anxiety exist to which it can be either considered as a qualitatively distinct subtype of social phobia or a quantitatively less severe form of a more impairing generalized social phobia. However, the prevalence of public speaking fears can be regarded as high and there is considerable evidence for interference with work or education. In addition, public speaking anxiety can cause marked distress suggesting that the impairment, at least in some individuals, is high enough to warrant professional treatment. Cognitive behavioral therapy (CBT) has turned out as an effective treatment for social phobia in general but also for public speaking anxiety. Nevertheless, some aspects hinder the successful delivery of CBT to anxious individuals. On the one hand, individuals are sometimes uncertain if the severity of their symptoms and impairment justifies professional treatment. On the other hand, groups are required for conducting exposure interventions.

This study tries to circumvent these limitations by lowering the access to treatment and by providing treatment in a group of anxious individuals. Large-group one-session treatments have been shown to be feasible in the treatment of specific phobias and fears and investigations revealed first evidence regarding their efficacy.

The COVID-19 pandemic makes it impossible to conduct face-to-face group sessions, so an online setting making use of a videoconference tool has been chosen.

In this study, the investigators plan to conduct an online large-group one-session treatment to reduce public speaking anxiety comprising different cognitive and behavioral techniques. First, anxiety and its function in general as well as factors causing, defining and maintaining public speaking anxiety are addressed in a psychoeducation phase. Second, different speaking tasks are conducted to expose the individuals to their feared situation on the one hand and to address common cognitive processes characterizing public speaking anxiety, e.g. self-focused attention, on the other hand. The exercises will be conducted in smaller groups.

Participants will be recruited from a community sample. They are invited to self-screen their public speaking anxiety to see if the intervention is suitable for them. The only exclusion criterion is not having the appropriate technical equipment for participation in a videoconference.

Public speaking anxiety as well as cognitive facets of social phobia will be assessed two months before treatment, two days before and one day after treatment and at one month and six months follow up to investigate long-term effects of the intervention.

Besides the aim of supporting a general feasibility and efficacy of the intervention, the study focusses on the role of expectancy violation. Recent theoretical frameworks suggest that expectancy violation is the core mechanism behind successful exposure therapy. Nevertheless, only a few studies to date manipulated expectancy violation experimentally to confirm its importance. Thus, participants in this study will be randomly allocated to two different treatment conditions. After completion of the treatment, one half of the participants will elaborate a worksheet that addresses basic contentual information concerning the treatment without a specific attempt to highlight the discrepancy between anticipated and actual outcomes. For example, participants will be asked how they would explain public speaking anxiety and exposure therapy to a friend and what advantages they see in conducting treatments like this in groups (BASIC task). The other group will receive a worksheet with questions aimed at enhancing the processing of what was learned during treatment in terms of expectancy violation. For example, they are asked if what they were most worried about occured and what actually happened compared to what they predicted to happen (EV task).

DETAILED DESCRIPTION:
Comprising both groups, the investigators expect a reduction in public speaking anxiety. This effect should be present comparing pre-treatment anxiety to the anxiety reported at the assessment points directly after treatment, one month after treatment and six months after treatment. The change in reported anxiety between the two assessment time points before treatment is used as a control condition as there is no waitlist control group that is assessed but not treated. The reduction in public speaking anxiety is expected to be larger when comparing the assessments before and after treatment than in the control period before treatment. Furthermore, the investigators hypothesize participants to benefit from the intervention in terms of other constructs, namely socially phobic cognitions and fear of negative evaluation.

Besides the hypotheses regarding general efficacy of the intervention, the investigators expect the reduction in public speaking anxiety in the EV group to be larger than in the BASIC group. This superiority of the EV condition should be present at the assessment points directly after treatment, one month after treatment and six months after treatment.

The sample under investigation will be a sample of anxious individuals recruited from the community. All participants can attain the intervention for free and there is no payment for participation. On a website created for the project, interested parties can receive information on the project and can self-screen their public speaking anxiety and generalized social anxiety. Participation is recommended if public speaking anxiety is high and if general social phobia is low. After registration for the study, participants are asked to fill out a survey through a link sent to them via e-mail. This survey comprises all outcome measures. The same procedure is carried out two days before, one day after, one month after and six months after treatment.

The target sample size is 100 participants. The decision for that number is not based on power calculations as there was no study before that conducted an online large-group one-session intervention for the treatment of public speaking anxiety and therefore effect size estimates would be random. Instead, the target sample size can be ascribed to organizational purposes.

In terms of the general efficacy hypothesis, the primary outcome measure will be analyzed with a repeated measures ANOVA covering the assessment time points after registration, two days before and one month after treatment.

For all other outcome measures, the investigators will use a rmANOVA comprising all five assessment time points, i.e. after registration, two days before the intervention, one day after the intervention, one month after the intervention and six months after the intervention. Furthermore, there will be paired comparisons between the public speaking anxiety scores at each of the assessment time points.

These analyses will be conducted not only for public speaking anxiety but also for social phobic cognitions, fear of negative evaluation and other psychological constructs such as positive mental health.

Regarding the expectancy violation hypothesis, the primary outcome measure will be analyzed with a 2x3 repeated measures ANOVA. For all other outcome measures, the investigators will use 2x5 between-within repeated measures ANOVAs (rmANOVA) to analyze the results. The first factor is a between-subjects factor that comprises the two groups BASIC and EV. The second factor is a within-subjects factor reflecting the five assessment time points after registration for the study, two days before the intervention, one day after the intervention, one month after the intervention and six months after the intervention. This analysis will be conducted for public speaking anxiety, social phobic cognitions and fear of negative evaluation. Moreover, there will be paired comparisons between the two groups for each of the assessment time points.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or above
* participants self-screen their public speaking anxiety and generalized social anxiety; participation is recommended if public speaking anxiety is moderate to high and if generalized social anxiety is low (this criterion is not explicitly checked by the investigator as there is only a recommendation and participants can register even though they do not receive a recommendation for participation)

Exclusion Criteria:

* Not having the appropriate technical equipment for participation in a videoconference

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
change on self statements during public speaking scale (german version; Hofmann & Heinrichs, 2001) | two days before the intervention and one month after the intervention [compared to the change between the assessment time points after registration and two days before treatment]
  10 items, 6-point Likert scale (0 - 5), large change in a negative direction means better outcome

SECONDARY OUTCOMES:
change on self statements during public speaking scale (german version; Hofmann & Heinrichs, 2001) | after registration for the study, two days before the intervention, one day after the intervention, one month after the intervention (already specified as primary outcome measure), six months after the intervention
  10 items, 6-point Likert scale (0 - 5), large change in a negative direction means better outcome
change on social cognitions questionnaire (german version; Stangier, Heidenreich, Ehlers, & Clark, 1996) | after registration for the study, two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  22 items, two questions regarding each item; 1st: frequency of thoughts, 5-point Likert scale (1 - 5), large change in a negative direction means better outcome; 2nd: degree of confidence, that the content of the cognition is correct, 0-100, large change in a negative direction means better outcome
change on fear of negative evaluation scale short form (german version; Kemper, Lutz, & Neuser, 2011) | after registration for the study, two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  5 items, 4-point Likert scale (1 - 4), large change in a negative direction means better outcome

OTHER OUTCOMES:
change on positive mental health scale (german version; Lukat, Margraf, Lutz, van der Feld, & Becker, 2015) | after registration for the study, two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  9 items, 4-point Likert scale (1 - 4), large change in a positive direction means better outcome
change on generalized self efficacy scale (german version; Schwarzer & Jerusalem, 1999) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  10 items, 4-point Likert scale (1 - 4), large change in a positive direction means better outcome
change on satisfaction with life scale (german version; Glaesmer, Grande, Braehler, & Roth, 2011) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  5 items, 7-point Likert scale (1 - 7), large change in a positive direction means better outcome
change on self-efficacy in presentation and moderation skills scale, presentation subscale (german version; Ringeisen, Rohrmann, Bürgermeister, & Tibubos, 2019) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  8 items, 5-point Likert scale (1 - 5), large change in a positive direction means better outcome
change on Rosenberg self-esteem scale - revised (german version; Collani & Herzberg, 2003) | two days before the intervention, one day after the intervention, one month after the intervention, six months after the intervention
  10 items, 4-point Likert scale (1 - 4), large change in a positive direction means better outcome
change on depression anxiety stress scale (DASS-21; german version; Nilges & Essau, 2015) | two days before the intervention, one month after the intervention, six months after the intervention
  21 items, 4-point Likert scale (0 - 3), 3 subscales that are analyzed separately (depression, anxiety, stress), large change in a negative direction means better outcome

CONTACTS AND LOCATIONS:
Overall Officials: Svenja Schaumburg, M. Sc., Principal Investigator — Ruhr University of Bochum
Locations (1):
- Ruhr-University of Bochum, Bochum, Germany

IPD SHARING:
Plan to Share IPD: Yes
It is planned to make individual participant data available on publication of the associated study results, via a publically-available data repository such as Open Science Framework. Data made available will be the research data reported in the publication, with the exception of any data that could compromise participant anonymity.